CLINICAL TRIAL: NCT00607061
Title: Synthesis of Glutathione in Erythrocytes From Low Birth Weight Newborn Babies : Effect of Cysteine in Vitro
Brief Title: Synthesis of Glutathione From Low Birth Weight Newborn Babies
Acronym: glutathione
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 06/12-O
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Low Birth Weight
Keywords: Glutathione; Cysteine; Synthesis rate; Newborns; Low birth weight newborn babies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other): Full term newborn babies with gestational age > 37 weeks of amenorrhea and weight of birth > tenth percentile.
  Interventions: Procedure: Blood sample collection
- 2 (Other): Low birth weight newborn babies (gestational age < 32 weeks of amenorrhea and/or weight of birth < 1500 g and/or weight of birth < third percentile for their gestational age.
  Interventions: Procedure: Blood sample collection
- 3 (Other): Full term newborn babies (gestational age > 37 weeks of amenorrhea and weight of birth > tenth percentile).
  Interventions: Procedure: Blood sample collection

INTERVENTIONS:
Procedure: Blood sample collection — Blood of the umbilical cord will be collected after delivery. A mother blood sample will be also collected in the few hours preceding delivery to determine glutathione and cysteine concentrations.

SUMMARY:
The aim of the study is to determine mechanisms leading to glutathione deficiency in low birth weight newborn babies. Compared to full term neonates, depletion in this population may be due to a decreased synthesis rate or to an enhanced utilization or a combination of both mechanisms.The protocol is constituted of two steps. The objective of the first step is to quantify the blood concentration of glutathione in the artery and the vein of umbilical cord in full term newborn babies. Objectives of the second step are to determine if the glutathione synthesis rate, measured in vitro, is lower in erythrocytes collected from umbilical cord blood of low weight newborn babies compared to full term newborn babies. In this case, the next objective will be to determine if the adjunction of an excess of cysteine in vitro can restore the glutathione synthesis rate in these cells.

ELIGIBILITY:
Inclusion Criteria (first step):

* Full term newborn babies
* Gestational age > 37 weeks of amenorrhea and weight of birth > tenth percentile
* Eutocic delivery

Inclusion Criteria (second step):

* Low birth weight newborn babies (gestational age < 32 weeks of amenorrhea and/or weight of birth < 1500 g and/or weight of birth < third percentile for their gestational age)
* Full term newborn babies (gestational age > 37 weeks of amenorrhea and weight of birth > tenth percentile)

Exclusion criteria (first and second step):

* Mother diastolic blood pressure > 90 mmHg during pregnancy,
* pH < 7.2 at umbilical cord and/or difference in pH < 0,02 between arterial pH and venous pH
* Dystocic delivery
* Bacterial or viral maternofoetal infection
* Foetal malformation
* Foetal disease
* Taking N-acetyl-cystein or vitamines and antioxidant minerals by the mother for the last 24 hours

Max Age: 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2007-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The glutathione concentration in umbilical cord in full term newborn babies, the glutathione concentration in umbilical cord of low birth weight newborn babies and the effect of the adjunction of an excess of cysteine on the glutathione synthesis rate.

CONTACTS AND LOCATIONS:
Overall Officials: Alice KUSTER, Doctor, Principal Investigator — Nantes University Hospital; Norbert WINER, Doctor, Study Chair — Nantes University Hospital; Jean-Christophe ROZE, Professor, Study Chair — Nantes University Hospital; Dominique DARMAUN, Professor, Study Chair — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, Nantes, France

REFERENCES:
- [Derived] De Luca A, Kuster A, Tea I, Darmaun D, Roze JC, Robins R, Hankard R. Plasma amino acid pools in the umbilical cord artery show lower 15N natural isotope abundance relative to the maternal venous pools. Isotopes Environ Health Stud. 2021 Mar;57(1):3-10. doi: 10.1080/10256016.2020.1817914. Epub 2020 Sep 24. PMID 32972258